CLINICAL TRIAL: NCT06419010
Title: Use of Leukocyte- and Platelet-Rich Fibrin in the Surgical Treatment of Medication-related Osteonecrosis of the Jaw: a Randomized Controlled Trial
Brief Title: Leukocyte- and Platelet-Rich Fibrin in the Surgical Treatment of Medication-related Osteonecrosis of the Jaw
Acronym: PeRFOrMand
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC31/21/0165
Record Dates: First submitted 2024-04-29; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Osteonecrosis of the Jaw
Keywords: therapeutics; surgical; autologous platelet concentrates; Platelet-Rich Fibrin; PRF
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients will benefit from surgery with the use of L-PRF.
  Interventions: Procedure: Surgery with the use of L-PRF
- Control group (Other): Patients will benefit from standard surgical treatment.
  Interventions: Procedure: Standard surgery

INTERVENTIONS:
Procedure: Surgery with the use of L-PRF — The study protocol is the same as the standard surgery one but with additional use of L-PRF membranes
  Arms: Experimental group
Procedure: Standard surgery — The standard surgical treatment, taking place in the operating room under general anesthesia
  Arms: Control group

SUMMARY:
Medication-related osteonecrosis of the jaw (MRONJ) is a rare but serious side-effect of antiresorptive therapies used in the management of bone diseases, such as osteoporosis or bone metastases. A surgical management can lead to a resolution of the disease, but with perfectible results. For this purpose, the use of autologous platelet concentrates (APC) can be useful. With this study, researchers aim to demonstrate the efficacy of L-PRF (Leukocyte- and Platelet-Rich Fibrin) as an adjunct to the surgical treatment of MRONJ in terms of wound healing.

DETAILED DESCRIPTION:
Resulting in bone loss, infection, pain or discomfort, the presence of MRONJ decreases the quality of life of patients. There isn't any consensus about the treatment modalities for MRONJ, nor about its main goals. Traditionally, therapeutics only aimed to control and prevent the progression of the disease, but recent studies suggest that a whole resolution can currently be expected, especially from surgical therapies. These, when indicated, are not only intended for the removal of the pathological tissue, but above all for an hermetic mucosal healing, preventing secondary infection of the underlying bone.

The L-PRF (Leukocyte- and Platelet-Rich Fibrin) is a second-generation APC, produced in a strictly autologous way, by extemporaneous centrifugation of the patient's own blood. A fibrin clot, containing leukocytes and thrombocytes, is thereby isolated and transformed into membranes by compression. Their appliance to the surgical site allows a slow release of growth factors and cytokines with a positive effect on the revascularization of the wound.

Unfortunately, scientific evidence of their efficiencies is lacking. Therefore, a protocol of randomized clinical trial is proposed, aimed at evaluating the effect of the adjunction of APC to surgical procedures on the complete mucosal healing and thus the resolution of the MRONJ.

The control treatment strategy consists of the complete removal of the necrotic bone, in bleeding margins, followed by a tension-free and hermetic closure. In the test group, suturing will be preceded by the application of L-PRF membranes under the wound.

Patients will be followed for 6 months, during which the maintain of wound closure will be monitored. An evaluation of pain, health-related quality of life and oral health-related quality of life, will also be reported, such as the occurrence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* MRONJ requiring surgical treatment according to AAOMS criteria (stage 2 or 3; failure of first-line treatments; sequestration of a necrotic bone block), the resection of which needs general anesthesia;
* Affiliates or beneficiaries of a social security scheme.
* Having given free and informed written consent.

Exclusion Criteria:

* Presence of a maxillo-mandibular neoplastic lesion;
* Presence of several MRONJ lesions;
* History of cervico-facial radiotherapy;
* Contraindication to general anesthesia;
* Reduced life expectancy (estimated at less than 6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of the use of L-PRF during the surgical treatment of MRONJ, compared to surgical treatment alone, on complete mucosal healing. | 6 months postoperatively
  Proportion of subjects presenting complete mucosal healing, i.e. a return to stage 0 or the "at risk" stage of the AAOMS classification.

SECONDARY OUTCOMES:
MRONJ stage - Month 1 | 1 month postoperatively
  Evaluation and comparison between the 2 groups of the evolution of the MRONJ stage - (improvement, stability, worsening).
MRONJ stage - Month 3 | 3 months postoperatively
  Evaluation and comparison between the 2 groups of the evolution of the MRONJ stage - (improvement, stability, worsening).
MRONJ stage - Month 6 | 6 months postoperatively
  Evaluation and comparison between the 2 groups of the evolution of the MRONJ stage - (improvement, stability, worsening).
the postoperative pain - Month 1 | 1 month postoperatively
  Pain will be subjectively evaluated by the patients using a Numerical Scale, according to a score from 0 (absence of pain) to 10 (maximum pain imaginable).
the postoperative pain - Month 3 | 3 months postoperatively
  Pain will be subjectively evaluated by the patients using a Numerical Scale, according to a score from 0 (absence of pain) to 10 (maximum pain imaginable).
the postoperative pain - Month 6 | 6 months postoperatively
  Pain will be subjectively evaluated by the patients using a Numerical Scale, according to a score from 0 (absence of pain) to 10 (maximum pain imaginable).
health-related quality of life - Month 1 - World Health Organization Quality of Life WHOQOL-BREF | 1 month postoperatively
  Overall quality of life will be assessed by the WHOQOL-BREF questionnaire
health-related quality of life - Month 1 - OHIP-14 | 1 month postoperatively
  oral health-related quality of life will be assessed via the OHIP-14 questionnaire.
health-related quality of life - Month 3 WHOQOL-BREF | 3 months postoperatively
  Overall quality of life will be assessed by the WHOQOL-BREF questionnaire and oral health-related quality of life will be assessed via the OHIP-14 questionnaire.
health-related quality of life - Month 3 Oral health-related quality OHIP-14 | 3 months postoperatively
  Oral Health Impact Profile of life will be assessed via the Oral Health Impact Profile OHIP-14 questionnaire.
health-related quality of life - Month 6 WHOQOL-BREF | 6 months postoperatively
  Overall quality of life will be assessed by the WHOQOL-BREF questionnaire
health-related quality of life - Month 6 - OHIP-14 | 6 months postoperatively
  Oral health-related quality of life will be assessed via the OHIP-14 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Claire VILLEPINTE, MD, Principal Investigator — University Hospital, Toulouse
Locations (6):
- France (6):
  - University Hospital - Centre François-Xavier Michelet, Bordeaux
  - University Hospital - Groupe hospitalier Pellegrin, Bordeaux
  - University Hospital, Limoges
  - University Hospital Gui de CHAULIAC, Montpellier
  - University Hospital Pitié-Salpêtrière, Paris
  - University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No